CLINICAL TRIAL: NCT04032431
Title: The Effect of a Telerehabilitation Virtual Reality Intervention on Functional Upper Limb Activities in People With Multiple Sclerosis
Brief Title: Upper Limb Telerehabilitation With Virtual Reality in Multiple Sclerosis
Acronym: TEAMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Cagliari (Other)
Collaborators: Azienda Sanitaria Locale di Cagliari (Other); Tel Aviv University (Other)
Responsible Party: Principal Investigator, Massimiliano Pau, Associate Professor, Head of the, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Italy-Israel-2019
Record Dates: First submitted 2019-07-17; First posted 2019-07-25 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Multiple Sclerosis
Keywords: Rehabilitation; Virtual Reality; Upper limb; Neurorehabilitation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: This is a prospective, assessor blinded, parallel group pilot RCT that will be conducted at:
  1. The Sardinian Center for Diagnosis and Treatment of Multiple Sclerosis, Cagliari, Italy.
  2. The Multiple Sclerosis Center, Sheba Medical Center, Tel-Hashomer, Israel.
  Participants will be randomly assigned to one of the two intervention groups:
  1. Telerehab VR training;
  2. Conventional therapy
  The two interventions will be comparable in length (8-weeks), frequency (twice weekly) and session duration (50-60 min).
  Pre-intervention tests (T0) characterizing groups and obtaining baseline values of primary and secondary outcome measures will be performed one week±3 days prior to the intervention program.
  Within one week after completion of the intervention, post-intervention tests will be performed (T1). The same tests will be repeated after 1-month of follow-up (T2). During the follow-up period (T1-T2), patients will be instructed to continue their regular activities.
Who Masked: Outcomes Assessor
Masking Description: Physical therapists and bioengineers in charge of outcome assessment are not involved in study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehab VR intervention (Experimental): The telerehab VR intervention consists of a custom-made software running on a computer connected with a commercial VR device (i.e. Oculus Rift). PwMS will be requested to reproduce several ADLs from the three main areas of self-care, dressing and meal preparation. The user can physically see his/her hands within the virtual scenario and, during the exercise, the hand coordinates are continuously recorded. Thus, data on 3D trajectory, speed, accuracy on target placement and movement smoothness, will be accessible. They will be stored in the PC and also be remotely sent to the clinical center for further analysis/processing. Both target position and task complexity will define the exercise difficulty, which can be modified automatically, on the basis of the previous performance or manually modified by the user
  Interventions: Behavioral: Telerehab VR intervention
- Conventional therapy (Active Comparator): Conventional therapy will focus on task-related upper-limb treatments while in a sitting or prone position, representing the standard care in MS. Several manual techniques, therapy tools and objects of ADL will be allowed during treatment. No restrictions will be placed on the material used (ie, ADL, reaching and grasping material). Use of additional electrical or mechanical therapy devices (ie, support arm systems, splints) will be avoided. The interventions will be conducted on a one-on-one basis in the physiotherapy or occupational therapy department of each participating center. Training and therapy content will be tailored to each participant's preferences, the agreed movement aims and the motor function level of each MS patient.
  Interventions: Behavioral: Telerehab VR intervention

INTERVENTIONS:
Behavioral: Telerehab VR intervention — Training with VR system using software specifically designed to reproduce activities of daily living

SUMMARY:
This study aims to investigate the effectiveness of a home-based telerehabilitation program specifically designed for upper limbs, based on Virtual Reality (VR) in individuals affected by Multiple Sclerosis.

DETAILED DESCRIPTION:
Approximately 60% of people with multiple sclerosis (pwMS) suffer from upper limb dysfunction. The primary goal of this study is to implement a single-blind, randomized control trial (RCT) designed to compare the effectiveness of an 8-week home-based telerehab virtual reality (VR) program with conventional therapy in pwMS with manual dexterity difficulties. Secondary aims include; a) evaluating the impact of the programs on quality of life after the intervention and a follow up 1 month later; and b) evaluating the impact of the programs on adherence and satisfaction.

Methodology. Twenty-four pwMS will be recruited to participate in the study which will be conducted at two established MS Centers: (1) The Sardinian Center for Diagnosis and Treatment of Multiple Sclerosis, Binaghi Hospital, Cagliari, Italy; (2) The Multiple Sclerosis Center, Sheba Medical Center, Tel-Hashomer, Israel. Participants will complete a total of three assessments focusing on upper limb functions. Both groups will receive 16 training sessions focusing on functional upper limb activities. The home-based telerehab VR intervention will comprise a custom-made software program running on a private computer or laptop. pwMS will perform several activities of daily living (ADL) functions associated with self-care, dressing and meal preparation.

Conventional therapy will focus on task-related upper-limb treatments while in a sitting or prone position, indicative of the standard care in multiple sclerosis (MS). Following 8-weeks of training, participants will complete a further outcome assessment. The same tests will be conducted 1 month (as a follow-up) after completion of the intervention.

Potential scientific contribution. The outcomes of this study have tremendous potential to improve the quality of evidence and informed decisions of functional upper limb activities in pwMS. If comparable results are found between the treatments in improving upper limb outcomes, this would suggest that pwMS can choose the program that best meets their personal needs, e.g., financial concerns, transportation or accessibility issues. Secondly, this information can be used by healthcare providers and medical professionals in developing upper limb exercise programs that will most likely succeed in pwMS and will then be disseminated to neurologists and other medical providers.

Mode of cooperation and added value. The Italian group will be responsible for designing and implementing three new VR scenarios relating to functional activities of the upper limb. The new VR scenarios will be planned in conjunction with the Israeli group who will also play an active role in the quality assessment procedures of the developed elements. Both groups will participate equally in the pilot RCT. Roles include: recruitment and guidance of patients and therapists, implementing the telerehab VR system in the patient's home, assessment of outcome measures, data collection, analysis and interpretation of data and dissemination of the findings. An additional role of the Israeli team will be to prepare a user manual detailing how to use the system and providing clinical guidelines/recommendations for both the therapist and patient.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of MS according to the revised McDonald Criteria 2017;
2. aged 25-60 years old;
3. an Expanded Disability Status Scale score ≥6;
4. an ability to understand and execute simple instructions;
5. a cut-off score of >0.5 pegs/s(=18s) on the NHPT (selected due to its high discriminative and predictive ability in distinguishing ADL independence in pwMS).

Exclusion Criteria:

1. orthopedic and other neurological disorders affecting upper limb movements (e.g., epileptic seizures);
2. contra-indication to physical activity (e.g., heart failure, severe osteoporosis);
3. moderate or severe cognitive impairments as indicated by the Mini-Mental State Examination score <21;
4. pregnancy (self-reported);
5. severe uncorrected visual deficits;
6. MS clinical relapse or treatment with corticosteroid therapy within 90 days prior to enrollment;
7. started or stopped a disease-modifying therapy for MS within 90 days prior to enrollment;
8. patients who received a course of physical or occupational therapy (home, outpatient or inpatient) within the past 30 days;
9. other treatments that could influence the effects of the interventions

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Nine Hole Peg Test (9HPT) | Pre-intervention (T0, baseline), post-intervention (T1, +8 weeks from baseline)
  The NHPT was selected based on the widespread adoption and extensive data available. Furthermore, the NHPT is recommended as a gold standard for measuring manual dexterity in pwMS.31 The NHPT has excellent psychometric properties regarding reliability, discriminant, concurrent and ecological validity, can detect progression over time, is sensitive to treatment and as such, is recommended for inclusion in clinical trials. Briefly explained, the NHPT requires participants to repeatedly place nine pegs into nine holes, one at a time, as quickly as possible and then remove them from the holes. The total time needed to complete the task is then recorded. Two consecutive trials with the dominant hand are immediately followed by two consecutive trials with the non-dominant hand.

SECONDARY OUTCOMES:
Action Research Arm Test (ARAT) | Pre-intervention (T0, baseline), post-intervention (T1, +8 weeks from baseline), 1 month follow-up (T2, +12 weeks from baseline)
  The ARAT is a 19 item observational measure used by physical therapists and healthcare professionals to assess upper extremity performance in terms of coordination, dexterity and functioning in several neurologic conditions, including MS.32 Items comprising the ARAT are categorized into four subscales (grasp, grip, pinch and gross movement) and arranged in order of decreasing difficulty, with the most difficult task examined first, followed by the least difficult task. Task performance is rated on a 4-point scale, ranging from 0 (no movement) to 3 (movement performed normally).
Manual Ability Measure-36 (MAM-36) | Pre-intervention (T0, baseline), post-intervention (T1, +8 weeks from baseline), 1 month follow-up (T2, +12 weeks from baseline)
  The MAM-36 is a questionnaire based on perceived ease or difficulty that a person may experience when performing unilateral and bilateral ADL tasks. During a semi-structured interview, the subject is asked to rate 36 unilateral and bilateral ADL tasks using a 4-point scale. The score of the different tasks are summed up and transformed using a Rasch-derived conversion table. The MAM-36 has adequate psychometric properties and is recommended as an outcome measure for upper limb function in pwMS
Value of "Impression of change" parameter | Pre-intervention (T0, baseline), post-intervention (T1, +8 weeks from baseline), 1 month follow-up (T2, +12 weeks from baseline)
  A 7-point Likert-type global rating scale from both the patient and therapist's perspective will be applied. The question that will be asked will be: "Compared to before treatment, at present, how would you rate your/the participant's functional upper limb activities?" The responses will be rated as: 1= worse than ever, 2 = much worse, 3 = slightly worse, 4 = unchanged, 5 = slightly improved, 6 = much improved, 7= greatly improved.

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Cocco, PhD, Principal Investigator — University of Cagliari
Locations (2):
- The Multiple Sclerosis Center, Sheba Medical Center, Tel Litwinsky, Israel
- Laboratorio di Biomeccanica ed Ergonomia industriale - Università degli Studi di Cagliari, Monserrato, Cagliari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kalron A, Achiron A, Pau M, Cocco E. The effect of a telerehabilitation virtual reality intervention on functional upper limb activities in people with multiple sclerosis: a study protocol for the TEAMS pilot randomized controlled trial. Trials. 2020 Aug 12;21(1):713. doi: 10.1186/s13063-020-04650-2. PMID 32787896